CLINICAL TRIAL: NCT07122804
Title: The Relationship Between Hyperventilation Symptoms and Physical Performance in Obese Individuals: An Observational Study
Brief Title: Hyperventilation and Physical Performance in Obesity
Status: Recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Kubra Koce, Asst. Prof., Istinye University
Other Study IDs: 2025/230
Record Dates: First submitted 2025-08-08; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Obesity
Keywords: Hyperventilation symptoms; Respiratory function; Physical performance
MeSH Terms: conditions — Obesity; Respiratory Aspiration | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Individuals aged between 18 and 65 years, with a Body Mass Index (BMI) ≥ 30 kg/m², who have the ability to understand and respond to the questionnaires and tests used in the study.
  Interventions: Other: Assessment

INTERVENTIONS:
Other: Assessment — Within the scope of the study, without any intervention, data regarding the participants' hyperventilation symptoms and physical capacities will be evaluated.

SUMMARY:
Obesity has become a major public health concern worldwide due to its rapidly increasing prevalence. It is defined as an abnormal or excessive accumulation of body fat that may impair health. Obesity is associated not only with chronic conditions such as cardiovascular diseases, type 2 diabetes, osteoarthritis, and certain types of cancer, but also with impaired respiratory function.

Excess body mass can reduce the range of motion of the respiratory muscles, limit the mechanical function of the chest wall and diaphragm, and decrease the efficiency of ventilation. As a result, individuals with obesity often experience exertional shortness of breath, rapid breathing, and inadequate ventilation. These symptoms may be considered part of hyperventilation syndrome, which is characterized by altered respiratory control and influenced by both physiological and psychological factors.

Although some studies have reported the presence of hyperventilation symptoms in individuals with obesity, their impact on physical performance has not been adequately investigated. Hyperventilation can limit the ability to perform daily activities and may lead to fatigue, imbalance, and other problems that directly affect physical performance.

The aim of this study is to examine the relationship between hyperventilation symptoms and physical performance parameters in individuals with obesity. The findings are expected to contribute to a more comprehensive assessment of physical fitness in this population and to support the development of individualized physiotherapy interventions.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18 and 65 years of age
* Having a Body Mass Index of 30 kilograms per square meter or higher (diagnosis of obesity)
* Providing written informed consent by signing the informed volunteer consent form after receiving information about the study
* Having sufficient physical and cognitive ability to individually perform the test procedures
* Being able to read and understand the Turkish language

Exclusion Criteria:

* Having a diagnosis of acute or chronic cardiovascular, pulmonary, rheumatological, neurological, or orthopedic disease
* Having a history of psychiatric illness (such as major depression, schizophrenia, or bipolar disorder)
* Having undergone major surgical operation within the past six months
* Having a level of physical limitation that prevents independent performance of daily living activities
* Being pregnant or in the breastfeeding period
* Having language, attention, or communication disorders that would prevent the administration of the Nijmegen Questionnaire

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals aged 18-65 with a Body Mass Index (BMI) ≥ 30 kg/m²
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Nijmegen Questionnaire: | 4 weeks
  The Nijmegen Questionnaire is a 16-item self-reported scale used to assess the subjective symptoms of hyperventilation syndrome. Each item is scored between 0 and 4, and individuals with a total score of 23 or higher are considered to have a high risk of hyperventilation
Chest Circumference Measurement | 4 weeks
  This is a simple anthropometric measurement used to indirectly assess respiratory capacity. The chest circumference is measured with a measuring tape during maximum inspiration and maximum expiration, and the difference between the two values is calculated
Modified Borg Scale | 4 weeks
  The Modified Borg Scale is a subjective tool used to measure perceived exertion and shortness of breath. It is rated from 0 (no difficulty) to 10 (maximum difficulty). It is particularly preferred for evaluations before and after the Six-Minute Walk Test.
Six-Minute Walk Test | 4 weeks
  The Six-Minute Walk Test is a practical and reliable field test used to evaluate lower extremity aerobic capacity and endurance. The individual is asked to walk as quickly as possible for six minutes along a flat corridor, and the total distance covered is recorded
Timed Up and Go Test | 4 weeks
  The Timed Up and Go Test is a practical and valid performance test used to evaluate mobility, balance, and functional movement abilities. In this test, the participant stands up from a chair, walks three meters, turns around, walks back, and sits down again. The time is measured in seconds, with shorter times indicating better functional performance. The Timed Up and Go Test is widely used to identify fall risk and mobility limitations, especially in older adults
Thirty-Second Sit-to-Stand Test | 4 weeks
  The Thirty-Second Sit-to-Stand Test is a functional test used to assess lower extremity muscle endurance. The participant is asked to stand up from and sit down on a chair as many times as possible within thirty seconds, and the number of repetitions is recorded
Modified Plank Test | 4 weeks
  The Modified Plank Test is a simple and safe test used to evaluate core stability. The participant is asked to maintain a plank position, supported on the elbows and knees, for as long as possible. The duration is measured in seconds.

SECONDARY OUTCOMES:
Quality of Life Instrument for Obese Individuals | 4 weeks
  The Quality of Life Instrument for Obese Individuals is a self-reported scale developed to evaluate obesity-specific quality of life and to assess the multidimensional impact of weight on quality of life in obese individuals. It measures the effects on areas such as physical functioning, self-esteem, sexual life, public distress, and work life. The instrument consists of thirty-one items and five subscales. Participants rate each statement on a five-point Likert-type scale ranging from "strongly disagree" (1) to "strongly agree" (5). The Turkish validity and reliability study of the instrument was conducted in 2024.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided